CLINICAL TRIAL: NCT05873816
Title: Cerebral Protection in Transcatheter Aortic Valve Replacement: The PROTEMBO Trial
Brief Title: The PROTEMBO Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Protembis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIP_00250
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Severe Aortic Valve Stenosis
Keywords: TAVR; Cerebral embolic protection
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- ProtEmbo - Cerebral Embolic Protection (Experimental): Subjects will undergo TAVR following placement of the ProtEmbo cerebral embolic protection device.
  Interventions: Device: ProtEmbo - Cerebral Embolic Protection
- Sentinel - Cerebral Embolic Protection (Active Comparator): Subjects will undergo TAVR following placement of the Sentinel cerebral embolic protection device.
  Interventions: Device: Sentinel - Cerebral Embolic Protection
- Control Arm (No Intervention): Subjects will undergo TAVR without embolic protection.

INTERVENTIONS:
Device: ProtEmbo - Cerebral Embolic Protection — Subjects will undergo TAVR following placement of the ProtEmbo cerebral embolic protection device.
  Arms: ProtEmbo - Cerebral Embolic Protection
Device: Sentinel - Cerebral Embolic Protection — Subjects will undergo TAVR following placement of the Sentinel cerebral embolic protection device.
  Arms: Sentinel - Cerebral Embolic Protection

SUMMARY:
The goal of this prospective, multi-center, randomized, controlled study is to compare the safety and efficacy of the ProtEmbo Cerebral Embolic Protection device to a hybrid control (no embolic protection device ('No Device') and the Sentinel device) in subjects with severe symptomatic native aortic valve stenosis indicated undergoing a TAVR procedure.

DETAILED DESCRIPTION:
Subjects with severe symptomatic aortic stenosis undergoing TAVR will be able to participate. Participants will be randomized in a 2:1:1 fashion to either the ProtEmbo arm, the Sentinel arm, or the 'No device' arm.

Enrolled subjects will undergo an MRI at baseline and at 36 hours ±12 hours, to evaluate any new cerebral lesions. Enrolled subjects will be followed for 30 days.

The study aims to address:

* whether the occurrence of all Major Adverse Cardiac and Cerebrovascular Events (MACCE) at 30 days is comparable between the ProtEmbo group and the hybrid control group.
* whether the total new lesion volume in the brain assessed by diffusion weighted magnetic resonance images at 36 ±12 hours is comparable between the ProtEmbo group and the hybrid control group.

ELIGIBILITY:
Inclusion Criteria:

1. The heart team recommends transcatheter aortic valve replacement via femoral access consistent with the 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease.
2. The subject and the treating physician agree that the subject will undergo the scheduled pre procedural testing and return for all required post procedure follow up visits.
3. The subject is able to provide informed consent, has been informed of the nature of the trial, agrees to its provisions and has provided written informed consent as approved by the relevant regulatory authority of the respective clinical site.
4. Subject is a minimum of 18 years of age.

Exclusion Criteria:

General exclusion criteria:

1. Subject is a woman of child-bearing potential.
2. Arm anatomy/ vasculature precluding radial or brachial artery access.
3. Hemodialysis shunt, graft, or arterio-venous fistula involving the upper extremity vasculature.
4. Evidence of an acute myocardial infarction ≤ 1 month before the intended treatment.
5. Severe ventricular dysfunction with LVEF ≤25%.
6. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 10 days of the index procedure.
7. Blood dyscrasias as defined by clinically significant leukopenia (< 500 leukocytes / μL), acute anemia (Hgb < 8 g / dL), thrombocytopenia (< 80,000 platelets / μl), history of bleeding diathesis or coagulopathy.
8. Hemodynamic instability, or pressure dependence requiring pharmacological inotropic support or mechanical heart assistance.
9. Echocardiographic evidence of intracardiac or aortic mass, thrombus not adequately treated, or vegetation.
10. Active peptic ulcer or upper GI bleeding within the prior 6 months.
11. Contraindication for anticoagulant or antiplatelet therapy.
12. Renal insufficiency (creatinine > 3.0 mg / dL or GFR < 30) and / or renal replacement therapy at the time of screening and dialysis patients.
13. Current or planned treatment with any investigational drug or investigational device during the study follow-up period (30 days).
14. Balloon aortic valvuloplasty (BAV) within 30 days of the procedure.
15. Cardiogenic shock, hemodynamic instability, or severe hypotension (systolic blood pressure < 90 mm Hg) at the time of the index procedure.
16. Cardiovascular surgical or interventional procedure 10 days prior or planned during the TAVR procedure or during the 30-day study follow-up.
17. Patients with severe chronic obstructive pulmonary disease (COPD)

NOTE: Use of general anesthesia during TAVR may affect neurocognitive function shortly after the procedure. While not an exclusion criterion, it is recommended that general anesthesia not be used if possible.

Neurological exclusion criteria:

1. Cerebrovascular event including TIA within 6 months of the procedure.
2. Subject had active major psychiatric disease.
3. Subject has severe visual, auditory, or learning impairment and is unable to comprehend English or local language and therefore unable to be consented for the study.
4. Subjects with neurodegenerative or other progressive neurological disease or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.

Magnetic resonance imaging exclusion criteria:

1. Body Mass Index (BMI) precluding imaging in scanner.
2. Contraindications to MRI (subjects with any implantable temporary or permanent pacemaker or defibrillator, metal implants in field of view, metallic fragments, clips, or devices in the brain or eye before TAVR procedure).
3. High risk of complete AV block after TAVR, with the need of permanent pacemaker (e.g., subjects with pre-existing bifascicular block or complete right bundle branch block plus any degree of AV block).
4. Planned implantation of a pacemaker or defibrillator implantation within the first 3 days after TAVR.
5. Claustrophobia precluding MRI scanning.

Anatomical and CT exclusion criteria:

1. Excessive tortuosity in left subclavian artery (≥ 70° single kink or ≥ 50° in sequential kinks).
2. Excessive tortuosity in right vascular access vessels for Sentinel introduction.
3. Significant stenosis (≥ 70%), calcification, ectasia, dissection, occlusion, aneurysm, or severe peripheral arterial disease in left or right arm access vessels - in particular at or within 3 cm of the aortic ostia.
4. Left subclavian artery diameter is ≤ 4 mm.
5. Brachiocephalic artery at the site of Sentinel filter placement < 9 mm or > 15 mm.
6. Left common artery at the site of Sentinel filter placement < 6.5 mm or > 10 mm.
7. Symptomatic or asymptomatic severe (≥ 70%) occlusive carotid disease requiring concomitant CEA / stenting.
8. Inner diameter of aortic arch < 25 mm as measured in any position between ascending aorta and ostium of left subclavian artery.
9. Distance between the origin of left subclavian artery and valve plain of < 90 mm.
10. Common ostium of cerebral vessels, where all three vessels originate from one single ostium in the aortic arch.
11. Significant stenosis, ectasia, dissection, aneurysm, or atheroma (mobile or > 5 mm thick) in the ascending aorta or in the aortic arch.
12. Significant angulation of the proximal segment of the left subclavian or aortic arch angulation or abnormal anatomical conditions of the aorta (a Type 3 aortic arch is not a reason for exclusion).
13. Distance between the origin of brachiocephalic trunk and left subclavian artery of > 65 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
MACCE at 30 days | Up to Day 30 post procedure
  Occurrence of Major Adverse Cardiac and Cerebrovascular Events (MACCE) at 30 days defined as all-cause mortality, all stroke, life-threatening or disabling bleeding, major vascular complications, and acute kidney injury (stage 2 or 3) as defined by VARC-3.
Total new lesion volume | 36 ±12 hours post TAVR procedure
  Total new lesion volume (TNLV) in the brain assessed by diffusion weighted magnetic resonance imaging (DW-MRI) at 36 ±12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (20):
- United States (15):
  - Tucson Medical Center Health, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - BayCare Health System / Morton Plant Hospital, Clearwater, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University - St. Louis, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - State University of New York at Buffalo, Buffalo, New York
  - NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center / NYPH, New York, New York
  - Weill Medical College / Cornell University, New York, New York
  - University of Texas, Memorial Hermann Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (4):
  - Dresden Herzzentrum, Dresden
  - Lübeck Universitätsklinikum Schleswig-Holstein Campus, Lübeck
  - Trier Krankenhaus der Barmherzigen Brüder, Trier
  - Ulm Universitätsklinikum, Ulm
- Gdansk Uniwersyteckie Centrum Kliniczne, Gdansk, Poland